CLINICAL TRIAL: NCT05212558
Title: The Rationale of Applying Inspiratory/Expiratory Muscle Training Within the Same Respiratory Cycle in Children With Bronchial Asthma: A Placebo-controlled Randomized Clinical Trial
Brief Title: Coupled Inspiratory and Expiratory Muscle Training in Children With Bronchial Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0020/0061
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Bronchial Asthma
Keywords: Chronic Respiratory Diseases; Respiratory Therapy; Chest Physiotherapy; Pulmonary Functions; Asthma; Respiratory Muscle Training
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled, assessor-blinded clinical trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded to the treatment allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): This group received a conventional respiratory retraining program plus unloaded (placebo) respiratory muscle training
  Interventions: Other: Placebo respiratory muscle training
- Inspiratory muscle training group (Active Comparator): This group received a conventional respiratory retraining program plus inspiratory muscle training only
  Interventions: Other: Inspiratory muscle training
- Combined training group (Experimental): This group received a conventional respiratory retraining program plus inspiratory and expiratory muscle training in the same respiratory cycle.
  Interventions: Other: Combined inspiratory and expiratory muscle training

INTERVENTIONS:
Other: Placebo respiratory muscle training — Unloaded respiratory muscle training plus conventional respiratory exercises
  Arms: Placebo group
Other: Inspiratory muscle training — Inspiratory muscle training plus conventional respiratory exercises
  Arms: Inspiratory muscle training group
Other: Combined inspiratory and expiratory muscle training — Combined inspiratory and expiratory muscle training in the same respiratory cycle plus conventional respiratory exercises.
  Arms: Combined training group

SUMMARY:
This study was designed to assess the effect of inspiratory and expiratory muscle training in the same cycle on respiratory muscle strength, pulmonary functions, perception of asthma symptoms in children with bronchial asthma. Fifty-one children with bronchial asthma were randomly allocated to the unloaded respiratory muscle training (Placebo training group; n = 17), inspiratory muscle training alone (inspiratory muscle training group; n = 17), or combined inspiratory and expiratory muscle training in the same cycle (combined training group; n = 17). All groups were assessed for respiratory muscle strength, pulmonary functions, and asthma symptoms.

DETAILED DESCRIPTION:
Fifty-one children with bronchial asthma were recruited from King Khalid Hospital, Al-Kharj, Saudi Arabia. The study included children who had a confirmed diagnosis of bronchial asthma according to the Global Initiative for Asthma guidelines, aged 12-18 years, identified as being stable cases, had a baseline percent-predicted value of the peak expiratory flow rate of 60-80%, sustained stale doses of medications in the past three months. Children who had unstable asthma or exacerbated asthma symptoms, history of thoracic surgery, or cardiopulmonary comorbidities were excluded.

Outcome measures

1. Respiratory muscle strength: assessed by measuring the maximal inspiratory and expiratory pressure using an electronic respiratory pressure meter.
2. Pulmonary function: The forced vital capacity (FVC), forced expiratory volume in the first second of expiration (FEV1), and FEV1/FVC ratio, were measured in a pulmonary function test through a spirometry analyzer.
3. Control of asthma symptoms: Asthma symptoms were assessed using a translated version of the asthma control test.

All groups received the conventional respiratory re-training program, three times a week, for 12 weeks in succession. The placebo group additionally received unloaded respiratory muscle training, the inspiratory muscle training group received respiratory muscle training alone, and the combined group received combined inspiratory and expiratory muscle training in the same cycle. Interventions were conducted by a licensed physical therapist who had experience of more than 10 years of respiratory training.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of asthma according to Global Initiative of Asthma guidelines.
* Age between 12 and 18 years.
* Clinically stable asthma.
* Stable doses of medications in the last three months
* A percent-predicted value of the peak expiratory flow rate of 60-80%
* No activity limitation due to asthma

Exclusion Criteria:

* Unstable asthma
* Exacerbation of asthma symptoms
* History of thoracic surgery
* Cognitive/behavioral problems
* Cardiopulmonary co-morbidities

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2020-08-02 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength | 2 months
  Inspiratory muscle strength was assessed by measuring the maximal inspiratory pressure (reflects the strength of the diaphragm and other inspiratory muscles) using an electronic respiratory pressure meter, according to the American Thoracic Society and European Respiratory Society standards. The highest value of three acceptable trials was documented and used for the subsequent analysis. The percent predicted maximal inspiratory pressure values (%) were calculated and used for statistical analysis.
Expiratory muscle strength | 2 months
  Expiratory muscle strength was assessed by measuring the maximal expiratory pressure (reflects the strength of the abdominal muscles and other expiratory muscles) using an electronic respiratory pressure meter, according to the American Thoracic Society and European Respiratory Society standards. The highest value of three acceptable trials was documented and used for the subsequent analysis. The percent predicted maximal inspiratory pressure values (%) were calculated and used for statistical analysis.
Forced vital capacity | 2 months
  Forced vital capacity, which is the amount of air that each participant was able to forcibly exhale from his/her lungs after taking the deepest breath they can, was measured in a pulmonary function test with a spirometry analyzer and expressed as a percentage of predicted values (%). Three trials were allowed and the best results were recorded.
Forced expiratory volume in one second | 2 months
  Forced expiratory volume in one second, which is the volume of air exhaled in the first second during forced exhalation after a maximal inspiration, was measured in a pulmonary function test with a spirometry analyzer and expressed as a percentage of predicted values (%). Three trials were allowed and the best results were recorded.
Forced expiratory volume in one second / forced vital capacity | 2 months
  Forced expiratory volume in one second / forced vital capacity, is the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs.

SECONDARY OUTCOMES:
Asthma symptoms | 2 months
  A translated version of the asthma control test was used to assess the degree of control over asthma symptoms. The test is patient-administered consists of 5 items. Each item has five possible responses (1: not controlled and 5: completely controlled). the test score ranges from 5 (inadequate control) to 25 (optimal control).

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No